CLINICAL TRIAL: NCT03167047
Title: Post-operative Pain Relief for Paediatric Inguinal-Scrotal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Kumarvel Veerappan (Other)
Responsible Party: Sponsor-Investigator, Dr Kumarvel Veerappan, Consultant Paediatric Anaesthatist, Medway NHS Foundation Trust
Organization: Medway NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16/LO/1187
Record Dates: First submitted 2017-02-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block (Active Comparator): Caudal epidural given for post-operative pain relief. Dose used is 1.5ml/kg of weak Levo-Bupivacaine solution (0.125%).
  Patients will also receive standardised pain relief of paracetamol and fentanyl
  Interventions: Procedure: Caudal block; Drug: Standarising intraoperative pain relief
- Nerve block (Active Comparator): Peripheral nerve block given for post operative pain relief. Levo-Bupivacaine 0.25% 2mg/Kg given under ultrasound guidance.
  Patients will also receive standardised pain relief of paracetamol and fentanyl
  Interventions: Procedure: Nerve Block; Drug: Standarising intraoperative pain relief

INTERVENTIONS:
Procedure: Caudal block — Caudal epidural
  Arms: Caudal block
Procedure: Nerve Block — Peripheral nerve block
  Arms: Nerve block
Drug: Standarising intraoperative pain relief — All patients will receive a standarised dose of paracetamol 15mg/kg and fentanyl 2mcg/kg.

SUMMARY:
Two methods of pain control in children undergoing surgery on the groin and scrotum are caudal injection (a form of epidural) with local anaesthetic, and a regional nerve block (an injection of local anaesthetic around the nerves supplying the area). A pilot study at our hospital showed a significant decrease in post-operative pain and nausea and vomiting in these two methods when compared to intravenous morphine and local anaesthetic to the wound.

One potential side effect from caudal injections is temporarily decreased motor power in the legs due to the local anaesthetic - it is thought that this might be overcome using a more dilute solution of local anaesthetic along with clonidine. This study is to demonstrate that this method is as effective as the use of a regional nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing day case elective inguinal-scrotal surgery

Exclusion Criteria:

* Contraindication to technique
* Significant comorbidities
* Patient/parent refusal

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Discharge postoperatively (approximately 2-4 hours postoperatively)
  FLACC for preverbal children
Pain relief | Discharge postoperatively (approximately 2-4 hours postoperatively)
  VAS for verbal children

SECONDARY OUTCOMES:
Motor paresis assessed with the Bromage score | Discharge postoperatively (approximately 2-4 hours postoperatively)
  Bromage score

CONTACTS AND LOCATIONS:
Overall Officials: Kumarvel Veerappan, FRCA, Principal Investigator — Medway NHS Foundation Trust
Locations (1):
- Medway NHS Foundation Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided